CLINICAL TRIAL: NCT00112879
Title: Phase II Study of Arsenic Trioxide, Ascorbic Acid, Dexamethasone, and Thalidomide in Patients With Previously Untreated High-Risk or Relapsed or Refractory Multiple Myeloma
Brief Title: Arsenic Trioxide, Ascorbic Acid, Dexamethasone, and Thalidomide in Treating Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCF-IRB-7469; CDR0000428248 (Registry Identifier: PDQ (Physician Data Query)); CCF-IRB-5241; CCF-CTI-T12016
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; Refractory Plasma Cell Neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Arsenic Trioxide; Ascorbic Acid; Dexamethasone; Thalidomide; Biological Therapy; Drug Therapy

INTERVENTIONS:
Drug: arsenic trioxide
Drug: ascorbic acid
Drug: dexamethasone
Drug: thalidomide
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: biological therapy
Procedure: chemotherapy
Procedure: drug resistance inhibition
Procedure: growth factor antagonist therapy
Procedure: non-specific immune-modulator therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Giving arsenic trioxide together with ascorbic acid, dexamethasone, and thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving arsenic trioxide together with ascorbic acid, dexamethasone, and thalidomide work in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with previously untreated high-risk or relapsed or refractory multiple myeloma (MM) treated with arsenic trioxide, ascorbic acid, dexamethasone, and thalidomide.
* Determine the safety of this regimen in these patients.

Secondary

* Determine the duration of response, progression-free survival, and overall survival of patients with previously untreated high-risk MM treated with this regimen.

OUTLINE: This is an open-label study.

* Induction therapy: Patients receive arsenic trioxide IV over 1-4 hours and ascorbic acid IV over 15-30 minutes on days 1-5 in week 1 and then twice weekly in weeks 2-12; oral dexamethasone on days 1-4, 11-14, 29-32, 39-42, 57-60, and 67-70 (weeks 1, 2, 5, 6, 9, and 10); and oral thalidomide once daily in weeks 1-12.
* Consolidation therapy: Beginning 4 weeks after completion of induction therapy, patients receive arsenic trioxide and ascorbic acid as in induction therapy; oral dexamethasone on days 1-4, 29-32, and 57-60 (weeks 1, 5, and 9); and oral thalidomide once daily in weeks 1-12.
* Maintenance therapy: Beginning 4 weeks after completion of consolidation therapy, patients receive arsenic trioxide IV over 1-4 hours and ascorbic acid IV over 15-30 minutes on days 1, 8, 15, and 22. Treatment with arsenic trioxide and ascorbic acid repeats every 90 days (every 12 weeks). Patients also receive oral dexamethasone on days 1-4. Treatment with dexamethasone repeats every 28 days. Patients receive oral thalidomide once daily. Maintenance therapy continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 33-68 patients (15-34 with previously untreated high-risk multiple myeloma [MM] and 18-34 with relapsed or refractory MM) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM), meeting 1 of the following criteria:
* Previously untreated disease with poor prognosis, meeting 1 of the following criteria:
* Active disease with β2 microglobulin ≥ 5.5 mg/dL
* Inactive disease with peripheral plasma cells OR chromosome 13 or 14 abnormalities by fluorescent in situ hybridization
* Relapsed or refractory disease
* Measurable disease by serum and urine M-protein and/or measurable plasmacytoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2* NOTE: *ECOG 3 allowed for patients with bone pain due to MM

Life expectancy

* At least 3 months

Hematopoietic

* Platelet count ≥ 75,000/mm^3 unless plasma cells > 50% in bone marrow
* Any WBC allowed provided plasma cells > 50% in bone marrow

Hepatic

* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN

Renal

* Creatinine ≤ 6.0 mg/dL

Cardiovascular

* Absolute QT interval ≤ 460 msec with potassium ≥ 4.0 mEq/L AND magnesium ≥ 1.8 mg/dL
* No conduction defects
* No unstable angina
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No New York Heart Association class II-IV heart disease
* No other significant underlying cardiac dysfunction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study therapy
* No blood, ova, or sperm donation during study participation
* No history of grand mal seizures except infantile febrile seizures
* No pre-existing neurotoxicity or neuropathy ≥ grade 2
* No uncontrolled diabetes mellitus
* No active serious infection that cannot be controlled with antibiotics
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No other condition that would preclude study compliance or follow up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior thalidomide allowed (in patients with relapsed or refractory MM)
* No prior thalidomide in combination with arsenic trioxide
* Prior epoetin alfa allowed

Chemotherapy

* See Biologic therapy
* Prior arsenic trioxide allowed (for patients with relapsed or refractory MM)
* No concurrent cytotoxic chemotherapy
* No chemotherapy within 2 weeks after completion of study treatment

Endocrine therapy

* Prior steroid therapy allowed (for patients with relapsed or refractory MM)

Radiotherapy

* No concurrent broad-field radiotherapy

Surgery

* Not specified

Other

* Prior and concurrent bisphosphonates allowed
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States